

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

## Statistical Analysis Plan: Mock-up Tables

Version 2.0, 10-FEB-2020

**Protocol Number: V203-AD-EXT** 

An Extension Study of a Phase IIa study in Patients with Mild Alzheimer's Disease to Evaluate the Safety, Tolerability, Immunogenicity, and Efficacy of UBITh® AD Immunotherapeutic Vaccine (UB-311)

Protocol version: 1.1, 22JAN2018

Sponsor: United Neuroscience Ltd., Taiwan Branch (UNS Taiwan)

Version 2.0, 10-FEB-2020 Protocol No.: V203-AD-EXT



# Statistical Analysis Plan: Mock-up Tables and Figures UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### **Table of Contents**

| Statis | tical A | nalysis Plan: Mock-up Tables | 1 |
|---|---|---|---|
| Table | of Cor | ntents | 2 |
| 1 | Statist | ical Changes from Study Protocol | 4 |
| 1.1 | 1 | Incorrect Treatment Group Assignment | 4 |
| 1.2 | 2 , | Analysis Populations | 5 |
| 1.3 | | Primary Endpoints - Response Rate | |
| 1.4 | | Primary Endpoints - Analysis of Immunogenicity Variable | |
| 1.5 | | Treatment Tolerability and Compliance | |
| 1.6 | | Secondary and Exploratory Endpoints | |
| 1.7 | | Exploratory Endpoints - Correlation between Titers of anti-A6 antibody with anti-measles or anti-HB es and Memory T cell responses for UBITh® 1 and UBITh® 2 | |
| 2 | | col Version | |
| 3 | | ical Methodology | |
| <b>3.</b> 1 | | Data Handling | |
| | 3.1.1 | Definition of baseline values | |
| | 3.1.2<br>3.1.3 | Data handling for outliers | |
| | 3.1.3 | Data handling for missing data | |
| | 3.1.5 | Data handling for protocol deviation | |
| | 3.1.6 | Data handling for withdrawals, dropouts, lost to follow-up | |
| | 3.1.7 | Data handling for early termination reason | |
| | 3.1.8 | Data handling for Laboratory category | |
| | 3.1.9 | Data handling for Computerized Cognitive Test | 12 |
| | 3.1.10 | Data handling for Disease Duration | 12 |
| 3.2 | 2 | General Statistical Methodology | 12 |
| 4 | Mock- | up Tables and Figures | 13 |
| Note: | : | | 13 |
| 14 | TABLE | S and FIGURES | 16 |
| 14 | . 1 | DEMOGRAPHIC DATA AND BASELINE CHARACTERISTICS | 16 |
| | 14.1.1 | | |
| | 14.1.2 | | |
| | 14.1.3 | | |
| | 14.1.4 | Study Disease History | 18 |
| | 14.1.5 | Previous Medical and Surgery / Procedure History and Concurrent Disease | 19 |
| | 14.1.6 | | |
| | 14.1.7 | Study Drug Administration, Overall Treatment Tolerability and Compliance | 20 |
| 14 | .2 | EFFICACY DATA | 22 |
| | 14.2.1 | | |
| | 14.2.2 | e , | |
| | 14.2.3 | | |
| | 14.2.4 | | |
| | 14.2.5 | i e | |
| | 14.2.6 | , , | |
| | 14.2.7 | , | |
| | 14.2.8 | Volumetric Magnetic Resonance Imaging (vMRI) | 24 |



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

| 14.2.9 | Volumetric Magnetic Resonance Imaging (vMRI) – By Main Study Treatment Group | 25 |
|---|---|---|
| 14.2.10 | Neurodegenerative Biomarkers | |
| 14.2.11 | Neurodegenerative Biomarkers – By Main Study Treatment Group | |
| 14.2.12 | Anti-Measles Antibody (Measles IgG), Anti-HBV Surface Antibody (HBsAb) | |
| 14.2.13 | Memory T Cell Response Test For UbithR 1 | 26 |
| 14.2.14 | Memory T Cell Response Test For UbithR 1 – By Main Study Treatment Group | 26 |
| 14.3 SAF | ETY DATA | 28 |
| 14.3.1 | Treatment Emergent Adverse Events – Subject Based Analyses | |
| 14.3.2 | Neurological Examinations and Local Tolerability at Injection Site | 32 |
| 14.3.3 | Laboratory Assessment – Hematology | 33 |
| 14.3.4 | Laboratory Assessment – Biochemistry | |
| 14.3.5 | Laboratory Assessment – Inflammatory | |
| 14.3.6 | Physical Examination | 35 |
| 14.3.7 | Vital Signs and Body Weight | 36 |
| 14.3.8 | Electrocardiography (ECG, EKG) | 37 |
| 14.3.9 | Safety Magnetic Resonance Imaging (sMRI) | 38 |
| SAP Amendme | nt History: | 40 |
| Reference: | | 40 |

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 1 Statistical Changes from Study Protocol

The statistical analysis methods will follow study protocol version 1.1 (22JAN2018). Due to incorrect treatment assignment (detailed in Section 1.2), the study was terminated earlier than the planned schedule. Exceptions and clarifications are described below:

#### 1.1 Incorrect Treatment Group Assignment

There are 3 treatment groups in main study V203-AD, corresponding dosing regimen is listed as table below.

Clinical schematic diagram in main study - V203-AD

| Treatment Group in V203-AD | Screening | | Treatment | | | | | | Follow | /-up | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | S1 S2 | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | V11 | V12 | V13 |
| Week | <b>-</b> 6 ∼ <b>-</b> 1 | 1 | 5 | 13 | 17 | 25 | 29 | 37 | 41 | 49 | 53 | 61 | 65 | 79 |
| UB-311 7 doses | | $\uparrow$ | $\rightarrow$ | $\uparrow$ | | $\uparrow$ | | <b>→</b> | | $\uparrow$ | | $\uparrow$ | | |
| UB-311 5 doses | | <b>↑</b> | <b>↑</b> | <b>↑</b> | | ↑P | | <b>↑</b> | | ↑P | | <b>↑</b> | | |
| Placebo | | ↑P | ↑P | ↑P | | ↑P | | ↑P | | ↑P | | ↑P | | |

<sup>↑:</sup> UB-311 ↑P: placebo

According to protocol, the dosing regimen in extension study V203-AD-EXT should follow table below.

Clinical schematic diagram in extension study - V203-AD-EXT

| Treatment<br>Group in V203-<br>AD | Planned<br>Treatment Group<br>in V203-AD-EXT | Screening | | | Т | reatment | | | | Follow-<br>up |
|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | S1 | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 |
| Week | | <b>-</b> 6 ∼ <b>-</b> 1 | 1 | 5 | 13 | 25 | 49 | 73 | 97 | 109 |
| UB-311 7 doses | UB-311 3 doses | | <b>↑</b> | ↑P | ↑P | | 1 | | 1 | |
| UB-311 5 doses | UB-311 3 doses | | <b>↑</b> | ↑P | ↑P | | 1 | | 1 | |
| Placebo | UB-311 5 doses | | <b>↑</b> | <b>↑</b> | <b>↑</b> | | <b>↑</b> | | <b>↑</b> | |

<sup>1:</sup> UB-311 1P: placebo (no injection after treatment unblinding of main study V203-AD)

However, incorrect treatment group assignment occurred during V203-AD-EXT study, and summary is given as below.

| Subject 1 | Jumbor | Actual Treatment Group in V203-AD-EXT | | |
|---|---|---|---|---|
| Subject 1 | Nullioci | UB-311 1 dose | UB-3113 doses | Total |
| | UB-311 7 doses | 10 | 2* | 12 |
| Treatment Group in | UB-311 5 doses | 7 | 5* | 12 |
| V203-AD | Placebo | 8* | 2 | 10 |
| | Total | 25 | 9 | 34 |

<sup>\*:</sup> incorrect treatment group assignment

There are 15 subjects who administered wrong treatment. From sponsor's judgment, the wrong treatment assignment is significantly impacting the primary endpoint. Consequently, the project is decided to be terminated and all subjects should finish all assessments at early termination visit.

As the study was early terminated by sponsor, there will be some visits or some measurement in the mock table(s) without data and will not be presented in the final table(s).

<sup>†:</sup> In V203-AD study, the week no. counts from 0, yet counts from 1 in V203-AD-EXT study. In order to be consistent with V203-AD-EXT, week no. in V203-AD study here are added 1.

#### Statistical Analysis Plan: Mock-up Tables and Figures

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 1.2 Analysis Populations

Per-protocol (PP) defined in protocol is listed below.

Section 9.2.1 "Efficacy populations" of study protocol

Per-protocol (PP) population: subjects who receive all planned doses of the study drug, complete the treatment period, fulfil all entry criteria, and have no key protocol deviation.

According to protocol section 9.2 "Efficacy populations" that one condition of Per-protocol (PP) population is "*complete the treatment period*", however, there will be no PP subjects due to early termination of the study. All efficacy analyses will be analyzed based on Modified Intent-to-Treat population and the conclusion will be made on Modified Intent-to-Treat population.

#### 1.3 Primary Endpoints - Response Rate

Response rate defined in protocol is provided below.

Section 9.1.2 "Immunogenicity variables" of study protocol

The level of anti-Aβ antibodies is one of the primary endpoints and is assessed at Week 1 (V1), Week 5 (V2), Week 13 (V3), Week 49 (V5), Week 97 (V7) and Week 109 (V8). The one-sided 95% confidence interval (CI, right side) from all visits (V1 to V13) for subjects in Arm 3 (placebo group) of V203-AD study will be calculated as the threshold of response. Antibody responders will be defined as the subjects with serum antibody titer > response threshold at any visit after first injection of UB-311.

Since there was randomization error in this study and there are only 2 valid placebo subjects, the analysis of response rate will be omitted.

#### 1.4 Primary Endpoints - Analysis of Immunogenicity Variable

Analysis of immunogenicity variable defined in protocol is listed below.

Section 9.3.3 "Analysis of immunogenicity variable" of study protocol

Immunogenicity analyses will be performed on the mITT and PP populations. The change in antibody level will be analyzed by a repeated-measures mixed-effects model.

Section 9.3.4 "Analysis of efficacy variables" of study protocol

Efficacy analyses will be performed on the mITT and PP populations. Descriptive statistics will be provided for all continuous variables at the scheduled visits. Continuous variables with repeated measures will be analyzed using a mixed-effects model.

Due to incorrect assignment and early termination resulting in more treatment groups and fewer visits than planned in the protocol, the Repeated-Measures Mixed-Effects Model is no longer appropriate. Change from baseline of each post-treatment visit will be presented in descriptive statistics instead.

#### 1.5 Treatment Tolerability and Compliance

According to protocol section 9.3.2, treatment tolerability and compliance will be derived by formulas below:

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

Section 9.3.2 "Treatment tolerability and compliance" of study protocol

The overall treatment tolerability of UB-311 is defined as the percentage of number of administered doses divided by number of administered doses plus number of missed doses of subject(s) who drops out due to drug-related AE(s). It is calculated according to the following formula:

$$100\% \text{ x } (A+B_1+C+D) / (A+B_1+B_2+C+D)$$

where

A: number of administered doses of completers

B<sub>1</sub>: number of administered doses of subject(s) who drops out due to drug-related AE(s)

B<sub>2</sub>: number of missed doses of subject(s) who drops out due to drug-related AE(s)

C: number of administered doses of subject(s) who drops out due to drug-unrelated AE(s)

D: number of administered doses of subject(s) who drops out not due to AE(s)

The overall compliance is defined as the actual dose (UB-311 or placebo) of injection compared to the prescribed dose of treatment during the study. It is calculated according to the following formula:

100% x (Actual injection dose/Prescribed injection dose)

Due to study early termination, the description of treatment tolerability and compliance is modified as below:

The overall treatment tolerability of UB-311 is defined as the percentage of number of administered doses divided by number of administered doses plus number of missed doses of subject(s) who drops out due to drug-related AE(s). Due to early termination of this study, for the purpose of calculating tolerability, the completers are defined as the subjects who finished all required doses before study termination by sponsor or treatment unblinding of V203-AD for placebo. It is calculated according to the following formula:

$$100\% \text{ x } (A+B_1+C+D) / (A+B_1+B_2+C+D)$$

where

A: number of administered doses of completers

B<sub>1</sub>: number of administered doses of subject(s) who drops out due to drug-related AE(s)

B<sub>2</sub>: number of missed doses (up to treatment unblinding of main study for placebo or study termination by sponsor) of subject(s) who drops out due to drug-related AE(s)

C: number of administered doses of subject(s) who drops out due to drug-unrelated AE(s)

D: number of administered doses of subject(s) who drops out not due to AE(s)

The overall compliance is defined as the actual dose (UB-311 or placebo) of injection compared to the prescribed dose of treatment during the study. It is calculated according to the following formula:

100% x (Actual injection dose/Prescribed injection dose)

=100% x (actual injected doses of  $(A+B_1+C+D)$ ) / (prescribed injection doses of  $(A+B_1+B_3+C+D)$ )

where

B<sub>3</sub>: number of missed doses (up to treatment unblinding of main study for placebo or study termination by sponsor) with visit date

#### Statistical Analysis Plan: Mock-up Tables and Figures

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 1.6 Secondary and Exploratory Endpoints

Secondary endpoints described in the protocol is provided below.

The secondary endpoints are to measure the treatment effects of UB-311 on:

- The change in cognitive and global assessments, including:
  - Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog)
  - Mini-Mental State Exam (MMSE)
  - Clinical Dementia Rating-Sum of Boxes (CDR-SB)
  - Computerized cognitive tests
- The change from baseline of V203-AD study in amyloid deposition by 18F-AV-45 PET imaging;

Due to the incorrect treatment assignment and study early termination, this study is underpowered for analyses with secondary endpoints. Therefore, all secondary endpoints will be considered as exploratory and the definition of Modified Intent-to-Treat Population will be revised as "Have both baseline and at least one post-baseline assessment in any of the primary variables, irrespective of compliance with the study protocol and procedures".

Exploratory analysis described in protocol is provided below.

The changes in anti-A $\beta$  antibody levels, cognitive and global assessments, PET, qEEG, brain volume and cortical thickness and neurodegenerative biomarkers in blood will be compared between the 3 treatment groups from V203-AD study. If subjects agree to provide his/her remaining specimens from V203-AD for neurodegenerative biomarkers analysis, the data will be also compared from baseline in V203-AD study between 3 treatment groups.

Due to the incorrect treatment assignment and early termination, it is not appropriate to perform statistical tests on the change in anti-A $\beta$  antibody levels, cognitive and global assessments, PET, qEEG, brain volume and cortical thickness and neurodegenerative biomarkers in blood compared between treatment groups. Hence these analyses will be omitted but descriptive statistics will be presented.

Exploratory endpoints (qEEG and cortical thickness) with substantial amount of missing data/visit due to study early termination or data quality issue cannot provide longitudinal evaluations so they will be omitted from analyses. No data listing or statistical analysis will be included in the SAP except what collected in EDC for these two exploratory endpoints.

# 1.7 Exploratory Endpoints - Correlation between Titers of anti-Aβ antibody with anti-measles or anti-HBV antibodies and Memory T cell responses for UBITh® 1 and UBITh® 2.

The correlation between titers of anti-A $\beta$  antibody and anti-measles or anti-HBV antibodies as well as memory T cell response for UBITh<sup>®</sup> 1 and UBITh<sup>®</sup> 2 described in protocol is given as below.

Section 6.3.1.6 "The correlation between titers of anti-Aβ antibody and anti-measles or anti-HBV antibodies as well as memory T cell response for UBITh® 1 and UBITh® 2"

The titers of anti-measles and anti-HBV antibodies will be compared to the maximum titer of anti-A $\beta$  antibody in subjects to evaluate the possible correlation between the titers of anti-A $\beta$  antibody elicited by UB-311 and anti-measles or anti-HBV antibodies in subjects.



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

Memory T cell response for UBITh® 1 and UBITh® 2 will be compared with titers of antimeasles or anti-HBV antibodies and anti-A $\beta$  antibody.

All planned exploratory analyses described above will be omitted due to insufficient data causing by early termination.

Version 2.0, 10-FEB-2020 Protocol No.: V203-AD-EXT



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 2 Protocol Version

The first subject was screened on 10-AUG-2018, and the last subject was dismissed on 30-OCT-2019 due to early termination of the study. All applied protocol and CRF versions are listed as below.

| No. | <b>Protocol Version</b> | CRF Version | IRB Approval | TFDA Approval |
|---|---|---|---|---|
| 1 | 1.1, 22JAN2018 | 2.1, 26JAN2018 | TVGH: 05FEB2018<br>NTUH: 08MAY2018<br>LK-CGMH: 03APR2018<br>KS-CGMH: 03APR2018 | 14MAR2018 |

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 3 Statistical Methodology

#### 3.1 Data Handling

Unless specially defined in corresponding sections, the data handling will follow tips below.

#### 3.1.1 Definition of baseline values

The baseline value of each assessment will be the value assessed closest and prior to UB-311/Placebo injection at Visit 1.

#### 3.1.2 Data handling for outliers

No data handling on outliers will be done.

#### 3.1.3 Data handling for missing data

Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog): ADAS-Cog-13 Total Score

- The calculation of ADAS-Cog-13 from ADAS manual 2015 includes ADAS-Cog-11 total items and 2 subscale (Maze and Cancellation Tasks).
- If more than one of 13 items of ADAS-Cog are missing/NA, ADAS-Cog-13 total score will be set to missing.
- The imputed total score of ADAS-Cog-13 when there is only one item is missing due to non-cognitive reasons is presented in:

| Missing Question | Imputed Total formula |
|---------------------|--------------------------|
| Word Recall | Observed Total*(1+10/75) |
| Orientation | Observed total*(1+8/77) |
| Word Recognition | Observed total*(1+12/73) |
| Delayed Word Recall | Observed Total*(1+10/75) |

#### **Memory T Cell Response Test**

Negative control:

- If negative control has a too numerous too count (TNTC) value, also called "Off scale well", it means the data has a quality control issue and the data is set as missing.
- For missing data at Visit 3 and Visit 8(ET), Screening Visit(S1) data will be used for imputation.
- Assume the negative control 0 as 1 in the analysis of fold change from negative control for Antigen 10 ug/ml, Antigen 5 ug/ml, Antigen 2.5 ug/ml.

Other condition (Positive Control, Antigen - 10 ug/ml, Antigen - 5 ug/ml, Antigen - 2.5 ug/ml):

• For the value is "Off scale well" or "Out well value", using the max from each cytokine including all concentrations and positive control across all subjects and all visits for imputation in the analysis of fold change from negative control.

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 3.1.4 Data handling for retest data

For the Laboratory Assessment, the retest result will be used for analysis instead of the first result, even if the collection date of retest data is after the injection date. For subject 02013E, the retest LB data (item: Potassium (K+)) that the date of retest is after the injection date will be used for analysis instead of the first result and the retest reason is due to hemolysis.

#### 3.1.5 Data handling for protocol deviation

Protocol deviations will be identified through programmatic checks of study data, as well as manual methods including clinical and monitoring reports. Statistician will examine the data by program in at least following aspects to confirm the protocol deviation list. The final protocol deviation list and population definition will be logged using TWDM-F17 "Protocol Violation & Population" form.

- Non-mITT population criteria
- Procedures/visits not done
- Procedures/visits out of time window
- Other protocol non-compliance.

#### 3.1.6 Data handling for withdrawals, dropouts, lost to follow-up

No data handling on withdrawals, dropouts, loss to follow-up will be done.

Visit 8 is an early termination visit since no subject completed all treatment visits due to study early termination. Measurements of visit 8 not in its visit window will not be adjusted.

#### 3.1.7 Data handling for early termination reason

There are 32 early termination subjects due to the study was early terminated by sponsor, therefore the reasons for early termination will be consolidated as below.

| Original reason | Recoded reason |
|---|---|
| by sponsor decided to terminate the long - | |
| term extension study with UB-311 <study< td=""><td></td></study<> | |
| v203-AD-EXT | |
| Based on review of V203-AD-EXT study | |
| baseline data on disease severity, and the | |
| treatment assignment error issue | |
| significantly impacting a primary endpoint, | Early Termination by Sponsor. |
| Sponsor (United Neuroscience Ltd.) | |
| executive team has evaluated the UB-311 | |
| clinical development pipeline and decided to | |
| terminate the long-term extension study with | |
| UB-311 (Study V203-AD-EXT). | |
| Early Termination by Sponsor. | |

The original reason will be presented in Listing and recoded reason will presented in Table.

#### Statistical Analysis Plan: Mock-up Tables and Figures

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 3.1.8 Data handling for Laboratory category

#### **Neurodegenerative Biomarkers**

"Not detectable" and "not tested" values will be set as missing for descriptive analysis.

#### Virology

Original results with both numerical value and categorical value (Positive/ Negative/ Equivocal), only categorical values will be presented for descriptive analysis.

#### Others (Biochemistry/Inflammatory/Hematology)

Original results with both numerical value and string value "<" or ">" will be transformed to exact numeric value with standard unit for descriptive analysis.

#### 3.1.9 Data handling for Computerized Cognitive Test

- 1. If completion = 1, excluding the data from all descriptive statistics
- 2. If the baseline is missing, exclude the subject from descriptive statistics of change from baseline
- 3. If data missing with completion = 0 and integrity = 1, add footnote in listing and indicate these data are "no correct response".

#### 3.1.10 Data handling for Disease Duration

For subjects (03001E, 03005E and 03007E) without Alzheimer's Disease record in this study, PET scan date of The Second Stage Screening from V203-AD study will be used to impute the missing onset date of Alzheimer's Disease diagnosis and derive their disease durations. Therefore, the onset date of Alzheimer's Disease diagnosis of these three subjects will be missing in Listing but their disease durations will be derived in Listing and Table.

#### 3.2 General Statistical Methodology

Descriptive statistics will be provided for all endpoints.

Continuous variables will be summarized by reporting the number of observations, mean, standard deviation, median, interquartile range (IQR = third quartile (Q3) - first quartile (Q1)), Q1, Q3, minimum and maximum, by group and overall.

Categorical variables will be summarized using frequency tables showing the number and percentage of subjects within a particular category, by group and overall.

Number of subjects at each visit will be based on the data with visit date.

#### Statistical Analysis Plan: Mock-up Tables and Figures

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 4 Mock-up Tables and Figures

The Mock-up "TABLES and FIGURES" is planned according to ICH E3, in which relevant CSR section is 14. The words shadowed below are to be adjusted or repeated upon real data, or just for notification.

Columns {Label, Treatment Groups, Total, Difference (if necessary)} will be included in the table with the analyzed population specified. In the mock table below, only the Label with one treatment column were presented to show the descriptive statistics to be displayed in the final tabulation. Column 'Difference' denotes pairwise comparison statistics.

#### For column Treatment Groups:

- It will be treatment group in V203-AD main study and actual treatment group in V203-AD-EXT extension study for tabulation.
- Treatment group in V203-AD main study will be added, respectively, for some section of 14.2 tabulation.

#### Note:

(1) Site ID  $\overline{\mathbb{C}}$ :

| Site ID | Full Name |
|---------|--------------------------------------------------|
| 01 | Taipei Veterans General Hospital (TVGH) |
| 02 | National Taiwan University Hospital (NTUH) |
| 03 | Linkou Chang Gung Memorial Hospital (LK-CGMH) |
| 04 | Kaohsiung Chang Gung Memorial Hospital (KS-CGMH) |

(2) Treatment group in V203-AD main study (unblinded on 01-NOV-2018) and actual treatment group in V203-AD-EXT extension study:

M7E1: 7 UB-311 injections in main study and 1 UB-311 injections in extension study

M7E3: 7 UB-311 injections in main study and 3 UB-311 injections in extension study

M5E1: 5 UB-311 injections + 2 Placebo injections in main study and 1 UB-311 injections in extension study

M5E3: 5 UB-311 injections + 2 Placebo injections in main study and 3 UB-311 injections in extension study

M0E1: 7 Placebo injections in main study and 1 UB-311 injections in extension study

M0E3: 7 Placebo injections in main study and 3 UB-311 injections in extension study

(3) Treatment group in V203-AD main study and regardless of the treatment group in extension study:

M7: 7 UB-311 injections in main study

M5: 5 UB-311 injections + 2 Placebo injections in main study

M7+M5: Once receiving UB-311 injection in main study

M0: 7 Placebo injections in main study

#### (4) Population

Version 2.0, 10-FEB-2020

Protocol No.: V203-AD-EXT

- Safety population:
  - (1) All subjects exposed to at least one dose of the study drug, regardless of the amount of treatment administered.
- Modified Intent-to-Treat Population (mITT):
  - (1) All subjects who receive at least one dose of the study drug
  - (2) Have both baseline and at least one post-baseline assessment in any of the primary variables, irrespective of compliance with the study protocol and procedures
- (5) For Visit Name (in Tables and Figures) and Visit Code (in Subject Data Listing):In the study, no Visits 5~7 data is collected and V8(ET) means early termination only since there is no Visit 8.

| Visit No. | Visit Description | Visit Day | Visit Name | Visit Code |
|---|---|---|---|---|
| 0 | Screen (Day -42 to -1) | -42 | Visit 0 (Screening) | V0 (S) |

#### Statistical Analysis Plan: Mock-up Tables and Figures

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

| Visit No. | Visit Description | Visit Day | Visit Name | Visit Code |
|---|---|---|---|---|
| 1 | Day 1 | 1 | Visit 1 (Day 1) | V1 D01 |
| 2 | Week 5 ± 3 Days | 29 | Visit 2 (Week 5) | V2 W05 |
| 3 | Week 13 ± 3 Days | 85 | Visit 3 (Week 13) | V3 W13 |
| 4 | Week 25 ± 14 Days | 169 | Visit 4 (Week 25) | V4 W25 |
| 5 | Week 49 ± 14 Days | 337 | Visit 5 (Week 49) | V5 W49 |
| 6 | Week 73 ± 14 Days | 505 | Visit 6 (Week 73) | V6 W73 |
| 7 | Week 97 ± 14 Days | 673 | Visit 7 (Week 97) | V7 W97 |
| 8 | Early Termination (ET) | Varied | Visit 8 (ET) | V8 ET |

#### (6) Treatment Tolerability and Treatment Compliance

The overall treatment tolerability of UB-311 is defined as the percentage of number of administered doses divided by number of administered doses plus number of missed doses of subject(s) who drops out due to drug-related AE(s). It is calculated according to the following formula:

 $100\% \text{ x } (A+B_1+C+D) / (A+B_1+B_2+C+D)$ 

where

A: number of administered doses of completers

B<sub>1</sub>: number of administered doses of subject(s) who drops out due to drug-related AE(s)

B<sub>2</sub>: number of missed doses (up to treatment unblinding of main study for placebo or study termination

by sponsor) of subject(s) who drops out due to drug-related AE(s)

C: number of administered doses of subject(s) who drops out due to drug-unrelated AE(s)

D: number of administered doses of subject(s) who drops out not due to AE(s)

The overall compliance is defined as the actual dose (UB-311 or placebo) of injection compared to the prescribed dose of treatment during the study. It is calculated according to the following formula:

100% x (Actual injection dose/Prescribed injection dose)

=100% x (actual injected doses of (A+B<sub>1</sub>+C+D)) / (prescribed injection doses of (A+B<sub>1</sub>+B<sub>3</sub>+C+D))

where

B<sub>3</sub>: number of missed doses (up to treatment unblinding of main study for placebo or study termination by sponsor) with visit date

#### (7) Full term for 'Protocol Deviation Code':

| Code | Full Term |
|---|---|
| | <to added="" be="" data="" final="" in="" real="" tabulation="" upon=""></to> |

#### (8) Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog): ADAS-Cog-13 Total Score

- The calculation of ADAS-Cog-13 from ADAS manual 2015 includes ADAS-Cog-11 total items and 2 subscale (Maze and Cancellation Tasks).
- If more than one of 13 items of ADAS-Cog are missing/NA, ADAS-Cog-13 total score will be set to missing.
- The imputed total score of ADAS-Cog-13 when there is only one item is missing due to non-cognitive reasons is presented in:

| Missing Question | Imputed Total formula |
|---------------------|--------------------------|
| Word Recall | Observed Total*(1+10/75) |
| Orientation | Observed total*(1+8/77) |
| Word Recognition | Observed total*(1+12/73) |
| Delayed Word Recall | Observed Total*(1+10/75) |

#### (9) MMSE and CDR-SB

No imputation will be performed if there is a missing point in MMSE or CDR-SB and the total score of MMSE or CDR-SB will be treated as missing.

#### (10) Neurodegenerative Biomarkers

"Not detectable" and "not tested" values will be set as missing for descriptive analysis.

#### (11) Virology

Version 2.0, 10-FEB-2020

Protocol No.: V203-AD-EXT

Original results with both numerical value and categorical value (Positive/ Negative/ Equivocal), only categorical values will be presented for descriptive analysis.

#### Statistical Analysis Plan: Mock-up Tables and Figures

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

(12) Others Laboratory (Biochemistry/ Inflammatory/ Hematology)

Original results with both numerical value and string value "<" or ">" will be transformed to exact numeric value with standard unit for descriptive analysis.

- (13) Memory T Cell Response Test Missing data estimation Negative control:
  - If negative control has TNTC value (off scale well), it means the data has quality control issue and set as missing.
  - For missing data at Visit 3 and Visit 8(ET), Screening Visit(S1) data will be used for imputation in the analysis of fold change.
  - Assume the negative control 0 as 1 in the analysis of fold change from negative control for Antigen 10 ug/ml, Antigen 5 ug/ml, Antigen 2.5 ug/ml.

Other condition (Positive Control, Antigen - 10 ug/ml, Antigen - 5 ug/ml, Antigen- 2.5 ug/ml):

- For the value is Off scale well or Out well value (too numerous to count, TNTC), using the max from
  each cytokine including all concentrations and positive control across all subjects and all visits for
  imputation.
- (14) Memory T Cell Response Test Fold change values for each test and concentration (Antigen-2.5 ug/ml, Antigen 5 ug/ml, or Antigen 10 ug/ml)
  - Fold change values at each visit:

Fold change value at visit =  $\frac{\text{value at visit}}{\text{Negative Control value at visit}}$ 

• Fold change values for change from baseline:

Fold change value for change from baseline (visit – baseline)

= Fold change value at visit − Fold change value at baseline

- (15) Structural MRI defined in protocol used for safety endpoints will be named as safety MRI and used for efficacy endpoints will be named as volumetric MRI.
- (16) For clinical relevant

CS: abnormal and clinically significant LLN: lower limit of normal range NCS: abnormal but not clinically significant ULN: upper limit of normal range

(17) Abbreviations of statistics

N: number of non-missing values Median: median of values

Missing: number of missing values IQR: inter-quartile-range (IQR=Q3-Q1)

Mean: mean of values

SD: standard deviation of values

O1: 25% quartile of values

CI: confidence interval

Q3: 75% quartile of values

(18) Full term for Amyloid-related Imaging Abnormalities (ARIA):

| ·). | Tun term for finificia felatea maging fiorermanties (firth f). | |
|---|---|---|
| | Code | Full Term |
| | ARIA-E | Vasogenic Edema and/or Sulcal Effusion |
| | ARIA-H | Hemosiderin Deposits |
| | ADE | Acute Disseminated Encephalomyelitis |
| | ARWMC | Age-Related White Matter Changes |
| | Non-ARIA | IA Other Significant Non-ARIA Abnormal Finding |



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 14 TABLES AND FIGURES

#### 14.1 DEMOGRAPHIC DATA AND BASELINE CHARACTERISTICS

## **14.1.1** Screen Failures and Subject Disposition by Study Site Population: All Screened Subjects / Enrolled Subjects

| Characteristics | Study Site |
|---|---|
| .All Screened Subjects | |
| N | XXX |
| ~Enrolled Subjects | XXX (XXX.X%) |
| ~Screening Failures | XXX (XXX.X%) |
| ~INC1 | XXX (XXX.X%) |
| ~INC2 | XXX (XXX.X%) |
| ~INC3 | XXX (XXX.X%) |
| ~EXC1 | XXX (XXX.X%) |
| ~EXC2 | XXX (XXX.X%) |
| ~EXC3 | XXX (XXX.X%) |
| Ziret | 11111 (11111117) |
| Enrolled Subjects | |
| N | XXX |
| Safety | XXX (XXX.X%) |
| ~mITT | XXX (XXX.X%) |
| ~ < Reason 1> | XXX (XXX.X%) |
| ~ < Reason 2> | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| ~Non-mITT | XXX (XXX.X%) |
| Non-Safety | XXX (XXX.X%) |
| Treatment group in V203-AD main study of Enrolled Subjects | |
| N | XXX |
| M7 | XXX (XXX.X%) |
| M5 | XXX (XXX.X%) |
| M0 | XXX (XXX.X%) |
| Actual Treatment group in V203-AD-EXT extension study of | |
| Enrolled Subjects | |
| N | XXX |
| E1 | XXX (XXX.X%) |
| E3 | XXX (XXX.X%) |
| 20 | 11111 (1111111) |
| Treatment group in V203-AD main study and Actual Treatment | |
| group in V203-AD-EXT extension study of Enrolled Subjects | |
| N | XXX |
| M7E1 | XXX (XXX.X%) |
| M7E3 | XXX (XXX.X%) |
| M5E1 | XXX (XXX.X%) |
| M5E3 | XXX (XXX.X%) |
| M0E1 | XXX (XXX.X%) |
| M0E3 | XXX (XXX.X%) |
| Protocol Deviction of Familiad Subjects | |
| Protocol Deviation of Enrolled Subjects N | VVV |
| | XXX |
| ~ Major | XXX (XXX.X%) |
| ~ < Reason 1> | XXX (XXX.X%) |
| ~ < Reason 2> | XXX (XXX.X%) |
| <br>Minan | XXX (XXX.X%) |
| ~ Minor | XXX (XXX.X%) |



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

| Characteristics | Study Site |
|--------------------------|--------------|
| ~ <reason 1=""></reason> | XXX (XXX.X%) |
| ~ < Reason 2> | XXX (XXX.X%) |
| | XXX (XXX.X%) |

Enrolled subjects: subjects who are enrolled in the extension study.

## 14.1.2 Study Visits, Study Termination, Subject Disposition and Protocol Deviation

| Pop | ulation: | Safety | Popu | lation |
|-----|----------|--------|------|--------|
|-----|----------|--------|------|--------|

| Characteristics | Treatment Group |
|---|---|
| . Study Termination | |
| N | XXX |
| Study Completed | XXX (XXX.X%) |
| Not Completed | XXX (XXX.X%) |
| ~ Withdrew consent | XXX (XXX.X%) |
| ~ Protocol issue | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| . Study Duration [days] | |
| | XXX |
| N (Missing)<br>Mean (SD) | |
| Median (IQR) | XXX (XXX) |
| | XXX (XXX) |
| Q1~Q3<br>Min. Mon. | XXX~XXX |
| Min~Max | XXX~XXX |
| .Population | |
| N | XXX |
| ~mITT | XXX (XXX.X%) |
| ~ < Reason 1> | XXX (XXX.X%) |
| ~ < Reason 2> | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| ~Non-mITT | XXX (XXX.X%) |
| .Protocol Deviation (Multi-Selection) | |
| N | XXX |
| ~ Major | XXX (XXX.X%) |
| ~ <reason 1=""></reason> | XXX (XXX.X%) |
| ~ <reason 2=""></reason> | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| <br>∼ Minor | XXX (XXX.X%) |
| ~ (Reason 1) | XXX (XXX.X%) |
| ~ < Reason 2> | · |
| ~ \Reason 2> | XXX (XXX.X%) |
| <b></b> | XXX (XXX.X%) |
| . Study Visits Completed (Multi-Selection by Status & mITT) | |
| N | XXX |
| Visit 0 (Screening) | XXX (XXX.X%) |
| ~ mITT | XXX (XXX.X%) |
| Visit 1 (Day 1) | XXX (XXX.X%) |
| ~ mITT | XXX (XXX.X%) |
| Visit 2 (Week 5) | XXX (XXX.X%) |
| ~ mITT | XXX (XXX.X%) |
| Visit 3 (Week 13) | XXX (XXX.X%) |
| ~ mITT | XXX (XXX.X%) |
| | , |



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

| Characteristics | Treatment Group |
|-------------------|-----------------|
| Visit 4 (Week 25) | XXX (XXX.X%) |
| ~ mITT | XXX (XXX.X%) |
| Visit 5 (Week 49) | XXX (XXX.X%) |
| ~ mITT | XXX (XXX.X%) |
| Visit 6 (Week 73) | XXX (XXX.X%) |
| ~ mITT | XXX (XXX.X%) |
| Visit 7 (Week 97) | XXX (XXX.X%) |
| ~ mITT` | XXX (XXX.X%) |
| Visit 8 (ET) | XXX (XXX.X%) |
| ~ mITT | XXX (XXX.X%) |

Study Duration [days] = Date of Termination - Visit 0, or alternatively as the last visit date - Visit 0

#### 14.1.3 Demographic Data

Population: Safety Population

| Characteristics | Treatment Group |
|--------------------------------------------------|-------------------|
| Study Sites | |
| N (Missing) | XXX (XXX) |
| Site 01 TVGH | XXX (XXX.X%) |
| Site 02 NTUH | XXX (XXX.X%) |
| Site 03 LK-CGMH | XXX (XXX.X%) |
| Site 04 KS-CGMH | XXX (XXX.X%) |
| Variable, including Age [Y/O], Body Weight [kg], | Body Height [cm], |
| BMI [kg/m^2] | |
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |
| Gender | |
| N (Missing) | XXX (XXX) |
| Male | XXX (XXX.X%) |
| 1,1010 | |

Age  $[Y/O] = int((date\ of\ informed\ consent-year/month/01\ of\ birth)/365.25)$ BMI  $[Kg/m^2] = body\ weight\ [kg]\ /\ body\ height\ [m]^2$ 

#### 14.1.4 Study Disease History

Population: Safety Population

| Characteristics | Treatment Group |
|---------------------------|-----------------|
| Disease Duration [years], | |
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | $XXX\sim XXX$ |
| Min~Max | $XXX\sim XXX$ |

Disease Duration [years] =(date of informed consent – onset date of Alzheimer's Disease diagnosis)/365.25, missing day is estimated as 15, missing month is estimated as Jul-01 For missing Alzheimer's Disease onset date, the PET scan date of The Second Stage Screening from V203-AD study will be used

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

## 14.1.5 Previous Medical and Surgery /Procedure History and Concurrent Disease

| Concurrent Disease | |
|---------------------------------------------|-------------------|
| Population: Safety Population | |
| Characteristics | Treatment Group |
| .Previous Medical History (Multi-Selection) | |
| . By MedDRA SOC, Preferred Term | |
| N | XXX |
| At least one below [Event#:Subj#] | XXX: XXX (XXX.X%) |
| <meddra body="" system1=""></meddra> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX: XXX (XXX.X%) |
| <meddra body="" system2=""></meddra> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX: XXX (XXX.X%) |
| .Current Condition (Multi-Selection) | |
| . By MedDRA SOC, Preferred Term | |
| N | XXX |
| At least one below [Event#:Subj#] | XXX: XXX (XXX.X%) |
| <meddra body="" system1=""></meddra> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX: XXX (XXX.X%) |
| <meddra body="" system2=""></meddra> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX: XXX (XXX.X%) |

Previous Medical History lists the medical histories with start date < date of Visit 1 Current Condition lists the medical histories that are ongoing or with end date  $\ge$  date of screening visit Based on the Medical Dictionary for Regulatory Activities (MedDRA version 21.1)

#### 14.1.6 Concomitant and Previous Medications

Population: Safety Population

| Characteristics | Treatment Group |
|-------------------------------------------|-----------------|
| .Previous Medications (Multi-Selection) | |
| N | XXX |
| At least one below | XXX (XXX.X%) |
| ~ <atc 1="" 3="" class="" level=""></atc> | XXX (XXX.X%) |
| ~ <atc 1="" preferred="" term=""></atc> | XXX (XXX.X%) |
| ~ <atc 2="" preferred="" term=""></atc> | XXX (XXX.X%) |
| *** | ••• |
| ~ <atc 2="" 3="" class="" level=""></atc> | XXX (XXX.X%) |
| ~ <atc 1="" preferred="" term=""></atc> | XXX (XXX.X%) |
| ~ <atc 2="" preferred="" term=""></atc> | XXX (XXX.X%) |
| .Concomitant Medications(Multi-Selection) | |
| N | XXX |



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

| Characteristics | Treatment Group |
|-------------------------------------------|-----------------|
| At least one below | XXX (XXX.X%) |
| ~ <atc 1="" 3="" class="" level=""></atc> | XXX (XXX.X%) |
| ~ <atc 1="" preferred="" term=""></atc> | XXX (XXX.X%) |
| ~ <atc 2="" preferred="" term=""></atc> | XXX (XXX.X%) |
| ••• | ••• |
| ~ <atc 2="" 3="" class="" level=""></atc> | XXX (XXX.X%) |
| ~ <atc 1="" preferred="" term=""></atc> | XXX (XXX.X%) |
| ~ <atc 2="" preferred="" term=""></atc> | XXX (XXX.X%) |
| | ••• |

Previous Medications lists the medications with start date < date of Visit 1

Concomitant Medication lists the medications that are ongoing or with end date ≥ date of Day 1 Medications are classified using the World Health Organization Drug Dictionary (WHODRUG) Anatomical Therapeutic Chemical (ATC) Level 3 classes and Preferred Terms (WHODRUG version WHODrug Global B3-format September 1, 2019)

Note: as medication is recorded from 3 months prior to screening visit to end of study, above definition is equivalent with the definition in section 9.3.1.2 in protocol as below.

- Previous medications are those that the subject took within 3 months period prior to the Screening visit and prior to the first administration of UB-311 at Week 1 (V1).
- Concomitant medications are those that the subject continued or started on or after the first injection of the study drug up to the end of the study.

## 14.1.7 Study Drug Administration, Overall Treatment Tolerability and Compliance

| Comphance | |
|---|---|
| Population: Safety Population | |
| Characteristics | Treatment Group |
| Gap Period [weeks], | |
| Total UB-311 + Placebo Dose [injections], | |
| Total UB-311 Dose [injections], | |
| Total UB-311 Dose [µg] | |
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |
| Overall Treatment Tolerability [%] | XXX.X |
| Treatment Compliance [%] | XXX.X |
| Injection Status \\ | |
| Visit 1 (Day 1) | |
| Visit 2 (Week 5) | |
| Visit 3 (Week 13) | |
| Visit 5 (Week 49) | |
| Visit 7 (Week 97) | |
| N (Missing) | XXX (XXX) |
| UB-311 Injection Completed | XXX (XXX.X%) |
| UB-311 Injection Not Completed | XXX (XXX.X%) |
| Placebo Injection Completed | XXX (XXX.X%) |
| Placebo Injection Not Completed | XXX (XXX.X%) |
| Not Done | XXX (XXX.X%) |
| UB-311 Dose [µg] for UB-311/Placebo injected sub<br>Visit 1 (Day 1)<br>Visit 2 (Week 5) | jects \\ |



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

| Characteristics | Treatment Group |
|-------------------|-----------------|
| Visit 3 (Week 13) | |
| Visit 5 (Week 49) | |
| Visit 7 (Week 97) | |
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |

Gap Period (weeks) = (First Injection Date in V203-AD-EXT study - The Last Injection Date in V203-AD study)/7

UB-311 is 300 µg per 0.5 mL per vial.

Refer to Note of title page for formula of Overall Treatment Tolerability [%] and Treatment Compliance [%] For group 'M7E1', 'M5E1' and 'M0E1', dosing at V2 and V3 are placebo.

The missing values are due to the IP issue at Site 2 except for the value of M5E1 and M7E1 group at Visits 2 and 3.

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 14.2 EFFICACY DATA

#### 14.2.1 Immunogenicity

- 14.2.1.1 Anti- $A\beta_{1-28}$  Antibody [Log 10] by Visit
- 14.2.1.2 Anti-Aβ<sub>1-42</sub> Monomer Antibody [Log 10] by Visit
- 14.2.1.3 Anti-A $\beta_{1-42}$  Oligomer Antibody [Log 10] by Visit
- 14.2.1.4 Anti-Aβ<sub>1-28</sub> Antibody [raw scale] by Visit
- 14.2.1.5 Anti-Aβ<sub>1-42</sub> Monomer Antibody [raw scale] by Visit
- 14.2.1.6 Anti-Aβ<sub>1-42</sub> Oligomer Antibody [raw scale] by Visit

< For 14.2.1.4-14.2.1.6, Log10\_Mean will be added, footnote: Log10\_Mean = log10 (Mean) >

#### 14.2.2 Immunogenicity – By Main Study Treatment Group

- 14.2.2.1 Anti-Aβ<sub>1-28</sub> Antibody [Log 10] by Visit
- 14.2.2.2 Anti-Aβ<sub>1-42</sub> Monomer Antibody [Log 10] by Visit
- 14.2.2.3 Anti-Aβ<sub>1-42</sub> Oligomer Antibody [Log 10] by Visit
- 14.2.2.4 Anti-Aβ<sub>1-28</sub> Antibody [raw scale] by Visit
- 14.2.2.5 Anti-Aβ<sub>1-42</sub> Monomer Antibody [raw scale] by Visit
- 14.2.2.6 Anti-Aβ<sub>1-42</sub> Oligomer Antibody [raw scale] by Visit

< For 14.2.2.4-14.2.2.6, Log10 Mean will be added,

footnote: Log10 Mean = log10 (Mean) >

#### <Layout 1: For Continuous Efficacy Assessment>

Population: Modified Intent-to-Treat Population

| Characteristics | Treatment Group |
|--------------------------------------------|-----------------|
| Visit 1 (Day 1), Baseline | |
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | $XXX\sim XXX$ |
| Min~Max | XXX~XXX |
| .Visit: Visit 2 (Week 5), Visit 3 (Week 13 | ), Visit 5 |
| (Week 49), Visit 7 (Week 97), Visit 8 (ET | |
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | $XXX\sim XXX$ |
| Min~Max | XXX~XXX |
| Visit - Baseline | |
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |

#### Statistical Analysis Plan: Mock-up Tables and Figures

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 14.2.3 Rating Scales

14.2.3.1 Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog): ADAS-Cog-13 Total Score

<Use Layout 1; except

Visits will be Visit 5, Visit 8. Refer to Note in title page for detail instruction>

14.2.3.2 Clinical Dementia Rating (CDR) Sum of Boxes Score

<Use Layout 1; except

*Visits will be Visit 5, Visit 8.* >

14.2.3.3 Mini-Mental State Examination (MMSE) Score

<Use Layout 1; except

*Visits will be Visit 5, Visit 8.* >

#### 14.2.4 Rating Scales – By Main Study Treatment Group

- 14.2.4.1 Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog): ADAS-Cog-13
  Total Score
- 14.2.4.2 Clinical Dementia Rating (CDR) Sum of Boxes Score
- 14.2.4.3 Mini-Mental State Examination (MMSE) Score

#### **14.2.5** Computerized Cognitive Test

- 14.2.5.1 Computerized Cognitive Test Detection Test (DET) on Speed of Performance [log10 msec]
- 14.2.5.2 Cognitive Test Identification Test (IDN) on Speed of Performance [log10 msec]
- 14.2.5.3 Computerized Cognitive Test International Shopping List Test (ISL) on Correct Responses [count]
- 14.2.5.4 Computerized Cognitive Test International Shopping List Test Delayed Recall (ISRL) on Correct Responses [count]
- 14.2.5.5 Computerized Cognitive Test Modified Groton Maze Learning Test (GML) on Total Errors [count]
- 14.2.5.6 Computerized Cognitive Test One Back Test (ONB) on Speed of Performance [log10 msec]

< Use Layout 1; except

- 1. Visits will be Visit 4, Visit 5, Visit6, Visit 8.
- 2. Practice data will be excluded>

#### 14.2.6 <sup>18</sup>F-AV-45 PET - Mean Standard Uptake Value Ratio (SUVR)

#### 14.2.6.1 <sup>18</sup>F-AV-45 PET - Mean SUVR

Population: Modified Intent-to-Treat Population

| Characteristics | Treatment Group |
|-----------------------------|-----------------|
| .By Brain Region | |
| Baseline from V203-AD study | |
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |

Version 2.0, 10-FEB-2020 Protocol No.: V203-AD-EXT



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

| Characteristics | Treatment Group |
|---------------------------------|-----------------|
| .By Brain Region | - |
| Min~Max | XXX~XXX |
| Visit 7 (Week 97), Visit 8 (ET) | |
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | $XXX\sim XXX$ |
| Change form baseline | |
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |

Mean SUVR is calculated using Whole Cerebellum as Reference Region

| Brain Region |
|---------------------------|
| COMPOSITE_TARGET_WEIGHTED |
| FRONTAL_LOBE_L |
| FRONTAL_LOBE_R |
| TEMPORAL_LOBE_L |
| TEMPORAL_LOBE_R |
| PARIETAL_LOBE_PRECUNEUS_L |
| PARIETAL_LOBE_PRECUNEUS_R |
| OCCIPITAL_LOBE_L |
| OCCIPITAL_LOBE_R |
| CEREBELLAR_GRAY_MATTER |
| SUBCORTICAL_WHITE_MATTER |
| PONS |

## 14.2.7 <sup>18</sup>F-AV-45 PET - Mean Standard Uptake Value Ratio (SUVR) – By Main Study Treatment Group

14.2.7.1 <sup>18</sup>F-AV-45 PET - Mean SUVR

#### 14.2.8 Volumetric Magnetic Resonance Imaging (vMRI)

#### 14.2.8.1 Brain Volume

< Use Layout 1; except

1. Baseline will be Visit 0 (Screening), Visit will be Visit 3 and Visit 7

2. By Brain Region analyses will be presented>

| Brain Region |
|-------------------------|
| LEFT_HIPPOCAMPUS |
| RIGHT_HIPPOCAMPUS |
| TOTAL_HIPPOCAMPUS |
| LEFT_LATERAL_VENTRICLE |
| RIGHT_LATERAL_VENTRICLE |
| THIRD_VENTRICLE |
| FOURTH_VENTRICLE |

#### Statistical Analysis Plan: Mock-up Tables and Figures

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

| <b>-</b> |
|-----------------|
| TOTAL_VENTRICLE |
| WHOLE_BRAIN |

## 14.2.9 Volumetric Magnetic Resonance Imaging (vMRI) – By Main Study Treatment Group

14.2.9.1 Brain Volume

#### 14.2.10 Neurodegenerative Biomarkers

- 14.2.10.1 Neurodegenerative Biomarker Aβ<sub>1-40</sub> Peptide [pg/mL]
- 14.2.10.2 Neurodegenerative Biomarker Aβ<sub>1-42</sub> Peptide [pg/mL]
- 14.2.10.3 Neurodegenerative Biomarker Total tau [pg/mL]
- 14.2.10.4 Neurodegenerative Biomarker Neurofilament light chain [pg/mL]
- 14.2.10.5 Neurodegenerative Biomarker Phosphorylated neurofilament heavy chain [pg/mL]
- 14.2.10.6 Neurodegenerative Biomarker Glial fibrillary acidic protein [pg/mL]
- 14.2.10.7 Neurodegenerative Biomarker Ubiquitin C-terminal hydrolase L1 [pg/mL] < Use Layout 1; except
  Visits will be Visit 5, Visit 7, Visit 8.

footnote: "Not Detectable" and "Not Tested" values will be set as missing.>

#### 14.2.11 Neurodegenerative Biomarkers – By Main Study Treatment Group

- 14.2.11.1 Neurodegenerative Biomarker Aβ<sub>1-40</sub> Peptide [pg/mL]
- 14.2.11.2 Neurodegenerative Biomarker Aβ<sub>1-42</sub> Peptide [pg/mL]
- 14.2.11.3 Neurodegenerative Biomarker Total tau [pg/mL]
- 14.2.11.4 Neurodegenerative Biomarker Neurofilament light chain [pg/mL]
- 14.2.11.5 Neurodegenerative Biomarker Glial fibrillary acidic protein [pg/mL]

## 14.2.12 Anti-Measles Antibody (Measles IgG), Anti-HBV Surface Antibody (HBsAb)

14.2.12.1 Anti-Measles Antibody

#### 14.2.12.2 Anti-HBV Surface Antibody

Population: Modified Intent-to-Treat Population

| Characteristics | Treatment Group |
|---------------------------------|-----------------|
| Visit 0 (Screening), Baseline | |
| N (Missing) | XXX (XXX) |
| Positive | XXX (XXX) |
| Equivocal | XXX (XXX) |
| Negative | XXX (XXX) |
| Visit 3 (Week 13), Visit 8 (ET) | |
| N (Missing) | XXX (XXX) |
| Positive | XXX (XXX) |
| Equivocal | XXX (XXX) |

Version 2.0, 10-FEB-2020 Protocol No.: V203-AD-EXT

#### Statistical Analysis Plan: Mock-up Tables and Figures

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

| Characteristics | Treatment Group |
|---------------------------------|-----------------|
| Negative | XXX (XXX) |
| . Baseline to Visit | |
| N (Missing) | XXX (XXX) |
| Positive to Negative/ Equivocal | XXX (XXX) |
| Unchanged | XXX (XXX) |
| Negative/ Equivocal to Positive | XXX (XXX) |

#### 14.2.13 Memory T Cell Response Test For UbithR 1

- 14.2.13.1 Memory T Cell Responses (observed values) –Interferon gamma [Spot number]
- 14.2.13.2 Memory T Cell Responses (observed values) –Interleukin 2 [Spot number]
- 14.2.13.3 Memory T Cell Responses (observed values) –Tumor necrosis factor-alpha [Spot number]

<Observed values will be used>

< Use Layout 1; except

- 1. The tabulation will be separated by 5 levels {Negative Control, Positive Control, Antigen- 2.5 ug/ml, Antigen- 5 ug/ml, Antigen- 10 ug/ml}
- 2. Baseline will be Visit 0 (Screening),
- 3. Visits will be Visit 3 (Week 13), Visit 8 (ET).

#### footnote:

- 1. Normalized result of average will be used
- 2. Refer to Note of title pages for data handling rule >
- 14.2.13.4 Memory T Cell Responses (fold change values) Interferon gamma [Spot number]
- 14.2.13.5 Memory T Cell Responses (fold change values) Interleukin 2 [Spot number]
- 14.2.13.6 Memory T Cell Responses (fold change values) Tumor necrosis factoralpha [Spot number]
  - < 1. Fold change values from Negative Control will be used
  - 2. Assume Negative Control 0 as 1>

#### <Use Layout 1; except

- 1. The tabulation will be separated by 3 levels { Antigen- 2.5 ug/ml , Antigen 5 ug/ml, Antigen 10 ug/ml }
- 2. Baseline will be Visit 0 (Screening),
- 3. Visits will be Visit 3 (Week 13), Visit 8 (ET).

#### footnote:

- 1. Fold change value= Visit value / Negative Control value
- 2..Refer to Note of title pages for fold change values at each visit and fold change values for change from baseline>

## 14.2.14 Memory T Cell Response Test For UbithR 1 – By Main Study Treatment Group

- 14.2.14.1 Memory T Cell Responses (observed values) –Interferon gamma [Spot number]
- 14.2.14.2 Memory T Cell Responses (observed values) –Interleukin 2 [Spot number]

#### Statistical Analysis Plan: Mock-up Tables and Figures

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

- 14.2.14.3 Memory T Cell Responses (observed values) –Tumor necrosis factor-alpha [Spot number]
- 14.2.14.4 Memory T Cell Responses (fold change values) –Interferon gamma [Spot number]
- 14.2.14.5 Memory T Cell Responses (fold change values) –Interleukin 2 [Spot number]
- 14.2.14.6 Memory T Cell Responses (fold change values) –Tumor necrosis factor-alpha [Spot number]

Version 2.0, 10-FEB-2020 Protocol No.: V203-AD-EXT Confidential Page 27 of 40



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 14.3 SAFETY DATA

#### 14.3.1 Treatment Emergent Adverse Events – Subject Based Analyses

- 14.3.1.1 Treatment Emergent AEs Subjects with AEs by Intensity/Grade
- 14.3.1.2 Treatment Emergent AEs Subjects with AEs At Injection Site by Intensity/Grade

<Event # and subject # of Brain Microhemorrhages will be presented in this table if any.>

Population: Safety Population

| Characteristics | Treatment |
|-----------------------------------------------------|--------------------|
| -All sites, Site 1, Site 2, Site 3, Site 4 | |
| . By MedDRA SOC, Preferred Term, and Severity Grade | |
| N | XXX |
| At least one below [Event#:Subj#] | XXX: XXX (XXX.X%) |
| ~ <meddra body="" system1=""></meddra> | XXX : XXX (XXX.X%) |
| ~ <meddra 1="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| ~ Grade 1, Grade 2, Grade 3, Grade 4, Grade 5 | XXX : XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX: XXX (XXX.X%) |
| ~ Grade 1, Grade 2, Grade 3, Grade 4, Grade 5 | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX : XXX (XXX.X%) |
| ~ Grade 1, Grade 2, Grade 3, Grade 4, Grade 5 | XXX : XXX (XXX.X%) |
| ~ <meddra body="" system2=""></meddra> | XXX : XXX (XXX.X%) |
| ~ <meddra 1="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| ~ Grade 1, Grade 2, Grade 3, Grade 4, Grade 5 | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX : XXX (XXX.X%) |
| ~ Grade 1, Grade 2, Grade 3, Grade 4, Grade 5 | XXX : XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX : XXX (XXX.X%) |
| ~ Grade 1, Grade 2, Grade 3, Grade 4, Grade 5 | XXX : XXX (XXX.X%) |

For each MedDRA SOC or Preferred Term, Subject with multiple events are counted as one incidence. Based on the Medical Dictionary for Regulatory Activities (MedDRA version 21.1)

#### 14.3.1.3 Treatment Emergent AEs - Subjects with AEs - by Causality

## 14.3.1.4 Treatment Emergent AEs - Subjects with AEs At Injection Site - by Causality

<Event # and subject # of Brain Microhemorrhages will be presented in this table if any.>

Population: Safety Population

| Treatment |
|--------------------|
| XXX |
| XXX: XXX (XXX.X%) |
| XXX: XXX (XXX.X%) |
| XXX : XXX (XXX.X%) |
| XXX : XXX (XXX.X%) |
| XXX : XXX (XXX.X%) |
| XXX : XXX (XXX.X%) |
| XXX : XXX (XXX.X%) |
| XXX : XXX (XXX.X%) |



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

| Characteristics | Treatment |
|--------------------------------------------------|--------------------|
| -All sites, Site 1, Site 2, Site 3, Site 4 | |
| ~ <meddra body="" system2=""></meddra> | XXX : XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX:XXX(XXX.X%) |
| ~ Definitely Related, Probably Related, Possibly | XXX : XXX (XXX.X%) |
| Related, Unlikely, Unrelated | |
| ~ < MedDRA Preferred Term 2> | XXX: XXX (XXX.X%) |
| ~ Definitely Related, Probably Related, Possibly | XXX: XXX (XXX.X%) |
| Related, Unlikely, Unrelated | |
| ~ < MedDRA Preferred Term 3> | XXX: XXX (XXX.X%) |
| ~ Definitely Related, Probably Related, Possibly | XXX : XXX (XXX.X%) |
| Related, Unlikely, Unrelated | |

For each MedDRA SOC or Preferred Term, Subject with multiple events are counted as one incidence. Based on the Medical Dictionary for Regulatory Activities (MedDRA version 21.1)

#### 14.3.1.5 Treatment Emergent AEs - Subjects with Drug Related AEs

## 14.3.1.6 Treatment Emergent AEs - Subjects with Drug Related AEs At Injection Site

<Event # and subject # of Brain Microhemorrhages will be presented in this table if any.>

Population: Safety Population

| Characteristics | Treatment |
|--------------------------------------------|--------------------|
| -All sites, Site 1, Site 2, Site 3, Site 4 | |
| . By MedDRA SOC, Preferred Term | |
| N | XXX |
| At least one below [Event#:Subj#] | XXX: XXX (XXX.X%) |
| ~ <meddra body="" system1=""></meddra> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX : XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX : XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX : XXX (XXX.X%) |
| ~ <meddra body="" system2=""></meddra> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX : XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX : XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX: XXX (XXX.X%) |

For each MedDRA SOC or Preferred Term, Subject with multiple events are counted as one incidence. Based on the Medical Dictionary for Regulatory Activities (MedDRA version 21.1) Drug Related is defined as Definitely Related, Probable Related, or Possibly Related

#### 14.3.1.7 Treatment Emergent AEs - Subjects with Grade ≥3 AEs

## 14.3.1.8 Treatment Emergent AEs − Subjects with Grade ≥3 AEs At Injection Site <Event # and subject # of Brain Microhemorrhages will be presented in this table if any.>

Population: Safety Population

| Characteristics | Treatment |
|----------------------------------------------------|--------------------|
| -All sites, Site 1, Site 2, Site 3, Site 4 | |
| . By Severity Grade, MedDRA SOC and Preferred Term | |
| N | XXX |
| At least one below [Event#:Subj#] | XXX: XXX (XXX.X%) |
| ~ Grade ≥3, Grade 4, Grade 5 | XXX: XXX (XXX.X%) |
| ~ < MedDRA Body System 1> | XXX : XXX (XXX.X%) |
| | . , |

Version 2.0, 10-FEB-2020 Confidential United Neuroscience Ltd., Taiwan Branch
Protocol No.: V203-AD-EXT Page 29 of 40 (UNS Taiwan)
A2 Healthcare Taiwan Co.



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

| Characteristics | Treatment |
|--------------------------------------------------|--------------------|
| -All sites, Site 1, Site 2, Site 3, Site 4 | |
| ~ < MedDRA Preferred Term 1> | XXX : XXX (XXX.X%) |
| ~ Definitely Related, Probably Related, Possibly | XXX : XXX (XXX.X%) |
| Related, Unlikely, Unrelated | |
| ~ < MedDRA Preferred Term 2> | XXX : XXX (XXX.X%) |
| ~ Definitely Related, Probably Related, Possibly | XXX : XXX (XXX.X%) |
| Related, Unlikely, Unrelated | |
| ~ < MedDRA Preferred Term 3> | XXX : XXX (XXX.X%) |
| ~ Definitely Related, Probably Related, Possibly | XXX : XXX (XXX.X%) |
| Related, Unlikely, Unrelated | |
| ~ <meddra body="" system2=""></meddra> | XXX : XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX : XXX (XXX.X%) |
| ~ Definitely Related, Probably Related, Possibly | XXX : XXX (XXX.X%) |
| Related, Unlikely, Unrelated | |
| ~ < MedDRA Preferred Term 2> | XXX : XXX (XXX.X%) |
| ~ Definitely Related, Probably Related, Possibly | XXX : XXX (XXX.X%) |
| Related, Unlikely, Unrelated | |
| ~ < MedDRA Preferred Term 3> | XXX: XXX (XXX.X%) |
| ~ Definitely Related, Probably Related, Possibly | XXX : XXX (XXX.X%) |
| Related, Unlikely, Unrelated | |

Based on the Medical Dictionary for Regulatory Activities (MedDRA version 21.1)

#### 14.3.1.9 Treatment Emergent AEs - Action Taken with Study Medication

| Population: Safety Population | |
|---|---|
| Characteristics | Treatment |
| -All sites, Site 1, Site 2, Site 3, Site 4 | |
| . By Injection Site (At Injection Site + Not At Injection Site, | |
| At Injection Site, Not At Injection Site), Action Taken, | |
| MedDRA SOC and Preferred Term | |
| N | XXX |
| At least one below [Event#:Subj#] | XXX: XXX (XXX.X%) |
| ~ Drug interrupted / withdrawn, Drug interrupted, Drug | XXX : XXX (XXX.X%) |
| withdrawn | |
| ~ <meddra body="" system1=""></meddra> | XXX : XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX : XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX : XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX: XXX (XXX.X%) |
| ~ <meddra body="" system2=""></meddra> | XXX : XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX:XXX(XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX:XXX(XXX.X%) |

Based on the Medical Dictionary for Regulatory Activities (MedDRA version 21.1)



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### Treatment Emergent AEs – Subjects with SAEs 14.3.1.10

#### Treatment Emergent AEs - Subjects with SUSARs 14.3.1.11

SUSAR: Suspected Unexpected Serious Adverse Reaction (Unexpected **Treatment Related SAE)** 

| Characteristics |
|-----------------|
|-----------------|

Population: Safety Population

| Population: Safety Population | |
|---|---|
| Characteristics | Treatment |
| -All sites, Site 1, Site 2, Site 3, Site 4 for 14.3.1.10 | |
| -All sites for 14.3.1.11 | |
| By SAE Criteria, MedDRA SOC and Preferred Term, | |
| Causality, and Severity Grade | |
| N | XXX |
| At least one below [Event#:Subj#] | XXX: XXX (XXX.X%) |
| <sae criterion,="" criterion:="" either="" or<="" requires="" sae="" td=""><td>XXX: XXX (XXX.X%)</td></sae> | XXX: XXX (XXX.X%) |
| Prolongs Hospitalization, death, > | |
| <meddra body="" system1=""></meddra> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX: XXX (XXX.X%) |
| ~ Definitely Related, Probably Related, Possibly | XXX : XXX (XXX.X%) |
| Related, Unlikely, Unrelated | XXX : XXX (XXX.X%) |
| ~ Grade 1, Grade 2, Grade 3, Grade 4, Grade 5 | |
| ~ < MedDRA Preferred Term 2> | XXX : XXX (XXX.X%) |
| ~ Neuron Teleffed Telli 27 ~ Definitely Related, Probably Related, Possibly | XXX : XXX (XXX.X%) |
| Related, Unlikely, Unrelated | XXX : XXX (XXX.X%) |
| ~ Grade 1, Grade 2, Grade 3, Grade 4, Grade 5 | $AAA \cdot AAA (AAA.A/0)$ |
| Grade 1, Grade 2, Grade 3, Grade 4, Grade 3 | |
| ~ < MedDRA Preferred Term 3> | XXX:XXX(XXX.X%) |
| ~ Definitely Related, Probably Related, Possibly | XXX:XXX(XXX.X%) |
| Related, Unlikely, Unrelated | XXX : XXX (XXX.X%) |
| ~ Grade 1, Grade 2, Grade 3, Grade 4, Grade 5 | , |
| <meddra body="" system2=""></meddra> | XXX: XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX: XXX (XXX.X%) |
| ~ Definitely Related, Probably Related, Possibly | XXX: XXX (XXX.X%) |
| Related, Unlikely, Unrelated | XXX: XXX (XXX.X%) |
| ~ Grade 1, Grade 2, Grade 3, Grade 4, Grade 5 | |
| ~ <meddra 2="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| ~ Definitely Related, Probably Related, Possibly | XXX : XXX (XXX.X%) |
| Related, Unlikely, Unrelated | XXX : XXX (XXX.X%) |
| ~ Grade 1, Grade 2, Grade 3, Grade 4, Grade 5 | $AAA \cdot AAA (AAA.A / 0)$ |
| ~ Grade 1, Grade 2, Grade 3, Grade 4, Grade 3 | |
| ~ < MedDRA Preferred Term 3> | XXX:XXX(XXX.X%) |
| ~ Definitely Related, Probably Related, Possibly | XXX : XXX (XXX.X%) |
| Related, Unlikely, Unrelated | XXX : XXX (XXX.X%) |
| ~ Grade 1, Grade 2, Grade 3, Grade 4, Grade 5 | , |
| , | |

Based on the Medical Dictionary for Regulatory Activities (MedDRA version 21.1)



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 14.3.2 Neurological Examinations and Local Tolerability at Injection Site

#### 14.3.2.1 Neurological Examinations

Population: Safety Population
Characteristics
Treatment Group

#### Neurological Examination $\lor$

Visit 1 (Day 1) Visit 2 (Week 5)

Visit 3 (Week 13)

Visit 5 (Week 49)

Visit 7 (Week 97)

 N (Missing)
 XXX (XXX)

 Normal
 XXX (XX.X%)

 NCS
 XXX (XX.X%)

 CS (Medical History)
 XXX (XX.X%)

 CS (Adverse Event)
 XXX (XX.X%)

#### 14.3.2.2 Local Tolerability at Injection Site

Population: Safety Population

Characteristics Treatment Group

#### **Local Tolerability at Injection Site \**\

Visit 1 (Day 1)

Visit 2 (Week 5)

Visit 3 (Week 13)

Visit 5 (Week 49)

Visit 7 (Week 97)

N (Missing)XXX (XXX)TolerableXXX (XX.X%)Not tolerableXXX (XX.X%)Not doneXXX (XX.X%)

Version 2.0, 10-FEB-2020 Protocol No.: V203-AD-EXT

UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 14.3.3 Laboratory Assessment – Hematology

- 14.3.3.1 Hematology <Hematology Item 1 and Unit>
- 14.3.3.2 Hematology <Hematology Item 2 and Unit>
- 14.3.3.3 Hematology <Hematology Item 3 and Unit>
- 14.3.3.4 ...

#### 14.3.4 Laboratory Assessment – Biochemistry

- 14.3.4.1 Biochemistry < Biochemistry Item 1 and Unit>
- 14.3.4.2 Biochemistry <Biochemistry Item 2 and Unit>
- 14.3.4.3 Biochemistry < Biochemistry Item 3 and Unit>
- 14.3.4.4 ...

#### 14.3.5 Laboratory Assessment – Inflammatory

- 14.3.5.1 Inflammatory < Inflammatory Item 1 and Unit>
- 14.3.5.2 Inflammatory < Inflammatory Item 2 and Unit>
- 14.3.5.3 Inflammatory < Inflammatory Item 3 and Unit>
- 14.3.5.4 ...

#### <For continuous Laboratory Assessment – Hematology, Biochemistry and Inflammatory>

Population: Safety Population

| Characteristics | Treatment Group |
|---------------------------|-----------------|
| Visit 0 (Screening) | |
| Visit 1 (Day 1), Baseline | |
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |
| N (Missing) | XXX (XXX) |
| Normal | XXX (XX.X%) |
| NCS | XXX (XX.X%) |
| CS (Medical History) | XXX (XX.X%) |
| CS (Adverse Event) | XXX (XX.X%) |
| Visit 2 (Week 5) | |
| Visit 3 (Week 13) | |
| Visit 5 (Week 49) | |
| Visit 7 (Week 97) | |
| Visit 8 (ET) | |
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |
| N (Missing) | XXX (XXX) |
| Normal | XXX (XX.X%) |
| NCS | XXX (XX.X%) |
| CS (Medical History) | XXX (XX.X%) |
| CS (Adverse Event) | XXX (XX.X%) |



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

| Characteristics | Treatment Group |
|----------------------------------------|-----------------|
| Visit – Baseline, for all above visits | |
| except Visit 0 (Screening), Visit 1 | |
| (Day 1) and Baseline | |
| N (Missing) | XXX (XXX) |
| Relieved | XXX (XX.X%) |
| Unchanged | XXX (XX.X%) |
| Worsened | XXX (XX.X%) |

Improved: CS (Medical History or Adverse Event) at baseline to Normal / NCS at visit. Unchanged: including Normal at baseline to NCS at visit, NCS at baseline to Normal at visit. Worsened: Normal / NCS / CS (Medical History) at baseline to CS (Adverse Event) at visit



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 14.3.6 Physical Examination

#### 14.3.6.1 Physical Examination – All Abnormalities

Population: Safety Population

| Characteristics | Treatment Group |
|--------------------------------|-----------------|
| Visit 0 (Screening), | |
| Visit 1 (Day 1), | |
| Visit 2 (Week 5), | |
| Visit 3 (Week 13), | |
| Visit 4 (Week 25), | |
| Visit 5 (Week 49), | |
| Visit 6 (Week 73), | |
| Visit 7 (Week 97), | |
| Visit 8 (ET) | |
| N (Missing) | XXX (XXX) |
| At least one below | XXX (XXX.X%) |
| ~ <body 1="" system=""></body> | XXX (XXX.X%) |
| ~CS (Medical History) | XXX (XXX.X%) |
| ~CS (Adverse Event) | XXX (XXX.X%) |
| ~ <body 2="" system=""></body> | XXX (XXX.X%) |
| ~CS (Medical History) | XXX (XXX.X%) |
| ~CS (Adverse Event) | XXX (XXX.X%) |
| ~ <body 3="" system=""></body> | XXX (XXX.X%) |
| ~CS (Medical History) | XXX (XXX.X%) |
| ~CS (Adverse Event) | XXX (XXX.X%) |



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 14.3.7 Vital Signs and Body Weight

- 14.3.7.1 Vital Signs Temperature [degree C]
- 14.3.7.2 Vital Signs Respiratory Rate [breaths/min]
- 14.3.7.3 Vital Signs Systolic Blood Pressure [mmHg]
- 14.3.7.4 Vital Signs Diastolic Blood Pressure [mmHg]
- 14.3.7.5 Vital Signs Heart Rate [beats/min]
- 14.3.7.6 Vital Signs Weight [Kg]

Population: Safety Population

| Characteristics | Treatment Group |
|-----------------------------------------------|-----------------|
| Visit 0 (Screening) | |
| Visit 1 Day 1 (Pre-Dosing) | |
| Baseline | |
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |
| . Visit | |
| Visit 1 (Day 1, Post-Dosing) | |
| Visit 2 (Week 5, Pre-Dosing) | |
| Visit 2 (Week 5, Post-Dosing) | |
| Visit 3 (Week 13, Pre-Dosing) | |
| Visit 3 (Week 13, Post-Dosing) | |
| Visit 4 (Week 25) | |
| Visit 5 (Week 49, Pre-Dosing) | |
| Visit 5 (Week 49, Post-Dosing) | |
| Visit 6 (Week 73) | |
| Visit 7 (Week 97, Pre-Dosing) | |
| Visit 7 (Week 97, Post-Dosing) | |
| Visit 8 (ET) | |
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |
| Visit - Baseline, for all above visits except | |
| Visit 0 (Screening), Visit 1 Day 1 (Pre- | |
| Dosing) and Baseline | |
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |

Baseline is Visit 1 (Pre-Dosing) or alternatively as Visit 0 if Visit 1 (Pre-Dosing) data is not available.



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 14.3.8 Electrocardiography (ECG, EKG)

#### 14.3.8.1 Electrocardiogram - Overall Interpretation

Population: Safety Population

| Characteristics | Treatment Group |
|-------------------------------|-----------------|
| Visit 0 (Screening), Baseline | |
| N (Missing) | XXX (XXX) |
| Normal | XXX (XX.X%) |
| NCS | XXX (XX.X%) |
| CS (Medical History) | XXX (XX.X%) |
| CS (Adverse Event) | XXX (XX.X%) |
| Visit 5 (Week 49) | |
| Visit 8 (ET) | |
| N (Missing) | XXX (XXX) |
| Normal | XXX (XX.X%) |
| NCS | XXX (XX.X%) |
| CS (Medical History) | XXX(XX.X%) |
| CS (Adverse Event) | XXX (XX.X%) |
| Visit - Baseline | |
| N (Missing) | XXX (XXX) |
| Improved Unchanged | XXX (XX.X%) |
| Worsened | XXX (XX.X%) |
| | XXX (XX.X%) |

Improved: CS (Medical History or Adverse Event) at baseline to Normal / NCS at visit. Unchanged: including Normal at baseline to NCS at visit, NCS at baseline to Normal at visit. Worsened: Normal / NCS / CS (Medical History) at baseline to CS (Adverse Event) at visit



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### 14.3.9 Safety Magnetic Resonance Imaging (sMRI)

#### 14.3.9.1 sMRI - Overall Interpretation

Use the layout of ECG, where visit are Visit 3 (Week 13), Visit 7 (Week 97)>

#### 14.3.9.2 sMRI - Amyloid-related Imaging Abnormalities (ARIA) Types

| Ponu | lation | Safety | Popula | tion |
|------|--------|--------|--------|------|
| ronu | iauon. | Saletv | robula | ион |

| Treatment Group |
|-----------------|
| XXX (XXX) |
| XXX (XXX.X%) |
| VVV (VVV V0/) |
| XXX (XXX.X%) |
| XXX (XXX.X%) |
| VVV (VVV) |
| XXX (XXX) |
| XXX (XXX.X%) |
| XXX (XXX.X%) |



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

| Characteristics | Treatment Group |
|---|---|
| ~ARIA-E Parenchyma | XXX (XXX.X%) |
| ~ARIA-E Leptomeninges | XXX (XXX.X%) |
| ~ARIA-H (Hemosiderin Deposits) | XXX (XXX.X%) |
| ~ARIA-H Macrohemorrhages | XXX (XXX.X%) |
| ~ARIA-H Microhemorrhages | XXX (XXX.X%) |
| ~ARIA-H Superficial Siderosis | XXX (XXX.X%) |
| ~ADE (Acute Disseminated Encephalomyelitis Evidence) | XXX (XXX.X%) |
| ~ARWMC (Age-Related White Matter Changes Evidence) | XXX (XXX.X%) |
| ~Non-ARIA (Other Significant Non-<br>ARIA Abnormal Finding) | XXX (XXX.X%) |

New Findings: None at Visit 0 (Screening) to Observed at visit

Macrohemorrhages was classified under non-ARIA abnormal finding in V203-AD study and classified under ARIA-H in V203-AD-EXT study. There was no finding of macrohemorrhages in V203-AD-study



UB-311 Extension for Mild Alzheimer's Disease who participated in V203-AD trial

#### **SAP Amendment History:**

| | sion Date De | Version |
|---|---|---|
| | .0 16-DEC-2019 N/. | 1.0 |
| 4.2.1.6 and variable is Visit Visit Visit Visit Colerability | • | 2.0 |
| Vis<br>Vis<br>Vis<br>Tole | .0 10-FEB-2020 | 2.0 |

#### **Reference:**

1. Administration and Scoring Manual Alzheimer's Disease Assessment Scale – Cognitive (ADAS-cog)

